CLINICAL TRIAL: NCT02385695
Title: A Prospective Comparative Study to Evaluate Safety and Effectiveness of Dynamic Stabilization Versus Lumbar Fusion in Treatment of Multilevel Lumbar Disc Degeneration Disease
Brief Title: Study to Evaluate Safety and Effectiveness of Dynamic Stabilization Versus Lumbar Fusion in Treatment of Multilevel Lumbar Disc Degeneration Disease
Acronym: MLIDH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qiang Zhou, MD. PhD. (Other)
Responsible Party: Sponsor-Investigator, Qiang Zhou, MD. PhD., Deputy Chair of the Department of Orthopedics, Chair of the Department of Spine Surgical Group, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: Scientific Research 2015 (06)
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Lumbar Spine Disc Degeneration
Keywords: Disc Degeneration Disease; DDD; multilevel lumbar Disc Degeneration Disease
MeSH Terms: interventions — Fracture Fixation, Internal; Gene Fusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Posterior Dynamic Stabilization: Surgical treatment with posterior dynamic stabilization
  Interventions: Procedure: Posterior Dynamic Stabilization
- Internal Fixation and Fusion: Surgical treatment with internal fixation and fusion
  Interventions: Procedure: Internal Fixation and Fusion

INTERVENTIONS:
Procedure: Posterior Dynamic Stabilization
  Groups: Posterior Dynamic Stabilization
Procedure: Internal Fixation and Fusion
  Groups: Internal Fixation and Fusion

SUMMARY:
The purpose of this study is to compare outcomes of (i) surgical treatment with posterior dynamic stabilization and (ii) surgical treatment with internal fixation and fusion in patients with multilevel lumbar degenerative disk disease.

DETAILED DESCRIPTION:
Study aims are:

1. To evaluate superiority of Surgical treatment with posterior dynamic stabilization compared to Surgical treatment with internal fixation and fusion in lumbar range of motion;
2. To compare Surgical treatment with posterior dynamic stabilization compared to Surgical treatment with internal fixation and fusion in functional outcomes as measured by change in Oswestry Disability Index;
3. To compare radiological, clinical, patient-reported and, safety outcomes between the two surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age between 30 and 75 years inclusive
3. Radiographic evidence of multi-level lumbar disc degeneration disease
4. Scheduled for 2- or 3-level lumbar discectomy at levels from L1 to S1 with or without dynamic stabilization or fusion
5. Preoperative ODI ≥ 30%
6. Clinical symptoms consistent with diagnosis of lumbar DDD:

   * Radicular back or lower extremity pain and/or
   * Decreased muscular strength and/or
   * Abnormal sensation
7. Failed to gain adequate symptom relief from at least one month of adequate non-operative treatment

Exclusion Criteria:

1. Cauda equina syndrome
2. Patients with other lumbar conditions that will, in the opinion of the investigator, interfere with clinical outcomes (e.g. spinal structural deformities, spinal fractures, ankylosing spondylitis, spinal tuberculosis, spinal infection, spinal tumors, symptomatic cervical spinal disease)
3. Osteoporosis defined as T-score ≤ -3.5. BMD will be measured by DEXA performed on lumbar spine
4. Systemic infection such as AIDS and active hepatitis
5. Recent history (less than 3 years) of chemical substance dependency or significant psychosocial disturbance, which may impact the outcome or study participation
6. Participation in a clinical trial of investigational drug or device within the past 30 days

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of The Third Medical University/Southwest Hospital with multilevel lumbar degenerative disk disease.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2015-03; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Range of Motion in Lumbar Spine | 24 Months

SECONDARY OUTCOMES:
Change in Oswestry Disability Index | 24 Months

OTHER OUTCOMES:
Numeric Rating Scale for Back Pain | 24 Months
Numeric Rating Scale for Leg Pain | 24 Months
Range of Motion in Sagittal Plane at Each Operated Level | 24 Months
Radiographic Evaluations by Woodend Classification and Modic Changes on MRI | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhou, MD, PhD, Principal Investigator — Third Military Medical University
Locations (1):
- Third Military Medical University/Southwest Hospital, Chongqing, China